CLINICAL TRIAL: NCT00523107
Title: PG2 Treatment for Improving Fatigue Among Advanced Cancer Patients Under Standard Palliative Care
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP012
Record Dates: First submitted 2007-08-21; First posted 2007-08-30 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Fatigue
Keywords: Fatigue; Standard Palliative Care; PG2; QLQ-C30; Compassionate
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PG2 (Experimental): PG2 500 mg / 500 ml normal saline will be given t.i.w for 8 weeks.
  Interventions: Drug: PG2
- Placebo (Placebo Comparator): 500 ml normal saline will be given t.i.w 1-4 weeks, then PG2 500 mg / 500 ml normal saline will be given 5-8 weeks.
  Interventions: Drug: PG2; Drug: Placebo

INTERVENTIONS:
Drug: PG2 — PG2 500 mg / 500 ml normal saline t.i.w. per week
Drug: Placebo — 500 ml normal saline t.i.w. per week
  Arms: Placebo

SUMMARY:
The objective of this study is to conduct a trial in the spirit of providing as much as possible the benefit of PG2 treatment to eligible patients and to evaluate the efficacy and safety of PG2 for relieving fatigue among advanced cancer patients who are under standard palliative care (SPC) at hospice setting and have no further curative options available. Patient's fatigue status, to be measured by the Brief Fatigue Inventory-Taiwanese Form (BFI-T), will be the primary endpoint. The fatigue improvement response rate among patients between two study arms will then be compared as the basis for efficacy evaluation at the end of the first treatment cycle, and will be the primary endpoint. Other endpoints, the fatigue improvement response rate and the mean fatigue scores change from baseline among patients within and between cycles will be included in the secondary efficacy endpoints, and will be compared between two study arms. Patients' quality of sleep, appetite, pain, fatigue, nausea, vomiting and global quality of life (QoL) will be also measured by 11 questions (SS11) from EORTC QLQ-C30 for secondary endpoint evaluation. The other secondary endpoints include Karnofsky performance scores, and weight change and its related c-reactive protein level of the patients.

* BFI-T (Brief Fatigue Inventory - Taiwan) : The BFI is a 9-item self-administered questionnaire which was developed by MD Anderson Cancer Center offers assessing levels of fatigue. Subjects rate each item based on how they felt for the preceding week using a 1-10 numeric rating scale (10 being the most unfavorable response). The single construct of the BFI allows for the mean of the nine items to be the overall score. The score is categorized as mild (1-3), moderate (4-6), and severe (7-10). The scale is a reliable instrument that correlates highly with similar fatigue and performance status measures.

DETAILED DESCRIPTION:
This is a trial to evaluate use of PG2 for fatigue improvement in advanced cancer patients who are under standard palliative care at hospice setting and have no further curative options available. Only patients who give consent to participate in this study and meet all other inclusion and exclusion criteria will be eligible to enroll into this study. All patients will continue the standard palliative care (SPC) during this study.

The main aim of this trial is to compare improvement of patient's fatigue status between patients with or without PG2 treatment. Patient's fatigue status will be assessed by the Brief Fatigue Inventory-Taiwanese (BFI-T) Form. Each patient's fatigue improvement response will be defined as an improvement in the mean fatigue scores by at least 10% from baseline. Other quality of life parameters will be measured by the 11 questions (SS11) of the EORTC QLQ-C30 and by Karnofsky performance scale. Patient's weight change and its related c-reactive protein will be followed. There are two study arms in this trial: 1) the PG2 plus SPC arm; and 2) the Placebo plus SPC arm.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form
* ≧ 18 years old
* Have locally advanced or metastatic cancer or inoperable advanced cancer
* Under standard palliative care (SPC) at hospice setting and have no further curative options available
* BFI fatigue score ≧ 4
* Women with childbearing potential must use contraception
* Life expectancy of at least 3 months as determined by the investigator
* Willing and able to complete quality of life questionnaires

Exclusion Criteria:

* Pregnant or breast-feeding females
* Uncontrolled systemic disease such as active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus
* Take central nervous system stimulators such as Methylphenidate within last 30 days
* In other investigational drug trials within last 30 days
* Karnofsky performance scores < 30%
* Diagnosed as dying status

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The fatigue improvement response rate among patients between two study arms will be compared as the basis for efficacy evaluation at the end of the first treatment cycle. | within and between each cycle (4 weeks)

SECONDARY OUTCOMES:
The fatigue improvement response rate among patients within and between cycles (by BFI-T) | within and between cycles (4 weeks)
The fatigue improvement by multiple BFI-T score levels among patients between two study arms | within and between cycles (4 weeks)
The mean fatigue scores change from baseline among patients within and between cycles (by BFI-T) | within and between cycles (4 weeks)
Symptoms/Quality of Life Assessments: SS11 of EORTC QLQ-C30 includes eleven questions to assess the symptoms/QoL parameters: sleep, appetite, pain, fatigue, nausea, vomiting and global quality of life | within and between cycles (4 weeks)
Karnofsky performance score | within and between cycles (4 weeks)
Weight change and the related blood c-reactive protein level | within and between cycles (4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Yuen-Liang Lai, M.D., Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, New Taipei City, Taiwan